CLINICAL TRIAL: NCT06486064
Title: Evaluating the Potential of Probiotic Supplementation Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chi-Chang Huang (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chi-Chang Huang, Dean of Research and Development Office, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B032
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Sleep Disorder; Anxiety; Depression; Stress; Probiotics
MeSH Terms: conditions — Sleep Wake Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- probiotics (Experimental): heat-treated Limosilactobacillus fermentum PS150
  Interventions: Dietary Supplement: heat-treated Limosilactobacillus fermentum
- placebo (Placebo Comparator): microcrystalline cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: heat-treated Limosilactobacillus fermentum — one capsule daily for 8 weeks
  Other Names: HT-PS150
  Arms: probiotics
Dietary Supplement: Placebo — one capsule daily for 8 weeks
  Arms: placebo

SUMMARY:
This study aims to evaluate the feasibility of probiotics in improving sleep indicators through clinical human studies. Previous animal experiments have confirmed that Limosilactob acillus fermentum PS150 and heat-treated Lactobacillus fermentum HT-PS150 strains have the effect of improving sleep. 90 subjects will be recruited, 45 in each group. They will be given either HT-PS150 or placebo for 8 weeks and their blood, urine, saliva and questionnaire will be evaluated.

DETAILED DESCRIPTION:
The most important function of sleep is to restore physical energy lost after activities during the day, and to adjust and reorganize people's emotions, behavior, and cognitive memory. The average adult sleeps about 7 to 8 hours. Good sleep quality has a great impact on the performance of work and study during the day. If a person does not get enough sleep for a long time, it is easy to suffer from memory loss, emotional instability and other phenomena. It will also affect the operation of the immune system and easily lead to colds and illnesses. The following statements are often complained by sleep disorder patient: 1. Difficulty falling asleep. 2. Difficulty maintaining sleep, often waking up suddenly in the middle of sleep or having difficulty falling back to sleep once woken up. 3. Waking up too early and having trouble falling back to sleep. This study aims to evaluate the feasibility of probiotics in improving sleep indicators through clinical human studies. Previous animal experiments have confirmed that Limosilactob acillus fermentum PS150 and heat-treated Lactobacillus fermentum HT-PS150 strains have the effect of improving sleep.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 60 years old
* Pittsburgh Sleep Quality Scale score is greater than or equal to 5
* Insomnia Severity Scale (ISI less than 22 points)
* Subjects need to have a regular daily routine (no night shift work)

Exclusion Criteria:

* Have used antibiotics or probiotic products in powder, capsule or tablet form within one month
* Are taking drugs that may affect sleep (for example: sleeping pills, antipsychotic drugs, corticosteroids, antihistamines, stimulants, etc.) or undergoing hormonal treatment (including birth control pills)
* Those who are taking traditional Chinese medicine or western medicine to treat serious acute diseases
* Patients with uncontrolled high blood pressure or diabetes, a history of cancer, and mental illness
* Those with a diagnosis of other sleep disorders besides insomnia (narcolepsy, restless legs, sleep apnea, etc.)
* People who are allergic to probiotic products
* Pregnant or breastfeeding
* Alcohol, tobacco and coffee addicts
* Have carried out long-distance travel or work across time zones in the past month and the next two months
* Those who have participated in other interventional clinical studies in the past three months
* Those who are judged by the moderator to be unsuitable to participate in the research

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index, PSQI | From baseline to 8 weeks assessed
  The Pittsburgh Sleep Quality Index contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Insomnia severity index, ISI | From baseline to 8 weeks assessed
  The ISI is a 7-item patient-reported outcome measure (PROM) assessing the nature, severity, and impact of insomnia on a 5-point Likert scale to rate each item from 0 (no problem) to 4 (very severe problem).

SECONDARY OUTCOMES:
Total sleep time | From one week before baseline to 8 weeks assessed
  Compare the sleep times on the Fitbit
Change in Generalised Anxiety Disorder Assessment (GAD-7) | From baseline to 8 weeks assessed
  The Generalised Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day"
Change in Depression Score Patient Health Questionnaire (PHQ-9) | From baseline to 8 weeks assessed
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression: The PHQ-9 incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool.Depression Severity: 0- none, 1-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Validity has been assessed against an independent structured mental health professional (MHP) interview. PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression.
Change in The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16, QLESQ-16 | From baseline to 8 weeks assessed
  The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 is a valid, reliable self-report instrument for assessing quality of life. The minimum raw score on the Q-LES-Q-16 is 14, and the maximum score is 70, higher scores mean a better outcome.
Change in Visual Analogue Scale-GI (VAS-GI) | From baseline to 8 weeks assessed
  Visual Analogue Scale for GI symptoms, VAS-GI (visual analogue scale, VAS 0-10) was designed to measure the response of symptoms and well-being in patients after taking probiotics or placebo.
Patient Global Impression scales of Improvement rated by patient（PGI-C） | From baseline to 8 weeks assessed
  The PGIC consists of one item taken from the clinical global impression and adapted to the patient. The minimum total score possible is 1 and the maximum total score possible is 7. Higher values represent a worse outcome.
Change in Melatonin in both blood and saliva | From baseline to 8 weeks assessed
Change in Cortisol in both blood and saliva | From baseline to 8 weeks assessed
  Cortisol is a steroid hormone that is produced by the adrenal glands which sit on top of each kidney. When released into the bloodstream, cortisol can act on many different parts of the body and can help: body respond to stress or danger increase body's metabolism of glucose control blood pressure reduce inflammation. Cortisol is also needed for the fight or flight response which is a healthy, natural response to perceived threats. The amount of cortisol produced is highly regulated by body to ensure the balance is correct.
Change in Total Antioxidant Capacity , TAC | From baseline to 8 weeks assessed
  Levels of Total Antioxidant Capacity , TAC in serum
Change in GABA in both blood and saliva | From baseline to 8 weeks assessed
  GABA is known for producing a calming effect. It's thought to play a major role in controlling nerve cell hyperactivity associated with anxiety, stress and fear.
Change in Serotonin in both blood and saliva | From baseline to 8 weeks assessed
  Serotonin is a chemical that carries messages between nerve cells in the brain and throughout your body. Serotonin plays a key role in such body functions as mood, sleep, digestion, nausea, wound healing, bone health, blood clotting and sexual desire. Serotonin levels that are too low or too high can cause physical and psychological health problems.
Change in Orexin in both blood and saliva | From baseline to 8 weeks assessed
  Orexin
Change in 6 sulfatoxymelatonin in urine | From baseline to 8 weeks assessed
  6 sulfatoxymelatonin
Change in Norepinephrine in both blood and urine | From baseline to 8 weeks assessed
  Norepinephrine
Changes in Interleukin-6 (IL-6) in saliva | From baseline to 8 weeks assessed
  changes in IL-6 blood serum concentration levels in serum experimental group (in comparison to placebo control)
Change in Gut microbiome | From baseline to 8 weeks assessed
  The gut microbiome plays important roles in both the maintenance of health and the pathogenesis of disease. Stool will be examined before and after probiotics.
Sleep quality | From baseline to 8 weeks assessed
  Compare the sleep score recorded on the Fitbit

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Institute of Sports Science, National Taiwan Sport University, Taoyuan District, Taiwan